CLINICAL TRIAL: NCT04709068
Title: Risk Stratification and Early Alerting Regarding COVID-19 Hospitalization
Acronym: RiskSEARCH
Status: Terminated | Type: Observational
Why Stopped: recruitment and enrollment challenges due to fast-changing landscape of pandemic
Sponsor: Current Health (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00047371
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Results first posted 2021-08-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Covid19
Keywords: wearable; at-home
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- COVID19+
  Interventions: Device: Current Health

INTERVENTIONS:
Device: Current Health — wearable device and tablet used to collect health measures at home

SUMMARY:
The purpose of this research is to remotely monitor individuals who have tested positive for COVID-19 to learn more about progression and recovery from the disease. Individuals who test positive for COVID-19 will wear the Current Health wearable device continuously and answer a brief series of questions on Current Health tablet daily for up to 30 days. The health data will be used to develop predictive models of hospitalization risk.

ELIGIBILITY:
Inclusion Criteria:

* Living in the United States (contiguous states)
* Aged 21 years or older
* Able to provide documentation of +Polymerase Chain Reaction (PCR) or +antigen test for COVID-19 within the past 48 hours
* Self-reports that comfortable and willing to wear the wearable device and interact with a tablet-based interface daily
* Able to provide a next of kin/designated person who can be contacted in the event of hospitalization for follow up.

Exclusion Criteria:

* Under the age of 21
* Received a positive test result more than 48 hours prior to contacting study staff or has a pending test for COVID-19
* Cannot confirm a PCR or antigen positive test for COVID-19
* Is unable to read English
* Is unwilling to wear the device 24 hours/day except for showering/bathing or interact with a tablet-based interface for daily questionnaire
* Is unwilling or unable to provide baseline data required for entry into the study
* Is unable to provide a next of kin/designated person who can be contacted in the event of hospitalization for follow-up
* Heavy tattooing on both upper arms
* Known atrial fibrillation (permanent or paroxysmal)
* Has taken/is taking part in a COVID-19 vaccine or treatment trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wolfberg, MD, Principal Investigator — Current Health
Locations (1):
- Current Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: study information and eligibility for enrollment — https://community.currenthealth.com/covid19-study

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COVID19+
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | COVID19+
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Participant Compliance
Description: a percentage of the number of 15 minute windows with vital sign data compared to the number of 15 minute windows with the potential to have vital sign data. The 15 minute windows with the potential to have vital sign data was calculated based on the number of days the participant was enrolled in the study. There were multiple study endpoints; the number of days varied between 14-30 days.
Time Frame: up to 30 days
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | COVID19+
Number analyzed (Participants) | 8
percentage of time | 74 [60 to 83]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | COVID19+
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT04709068/Prot_SAP_ICF_000.pdf